CLINICAL TRIAL: NCT02992145
Title: Androgens Level in the Third Trimester of Pregnancy in Patients With Preeclampsia
Status: Completed | Type: Observational
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Ismail Ahmed Mohamed, Obstetrics and gynaecology resident, Ain Shams Maternity Hospital
Other Study IDs: AinShams MH 01
Record Dates: First submitted 2016-12-12; First posted 2016-12-14 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Case group: This group will include forty (40) preeclampt
- Control group: This group will include forty (40) normoten

SUMMARY:
This study aims to compare between androgens level (serum total and free testosterone) in women with preeclampsia and normal ones in the third trimester of pregnancy (28-40 weeks).

DETAILED DESCRIPTION:
Methodology:

All women in this study will be subjected to:

* All women are candidates for this study according to inclusion and exclusion criteria.
* History taking with special emphases on last menstrual period to determine the exact Gestational age.
* A reliable date is defined as the occurrence of regular menstrual cycles (28±7 days) in patients who have not taken oral contraceptives during the three months before conception and have no irregular bleeding.
* General and abdominal examination for each patient to determine those patients matching with the inclusion criteria.
* Preeclampsia refers to the new onset of hypertension (systolic blood pressure ≥140 mmHg ,or diastolic blood pressure≥ 90 mmHg ,or both, measured on two occasions > 6 hours apart) and either proteinuria or end organ dysfunction after 20 weeks of gestation in a previously normotensive woman.
* At Ain Shams University Hospitals, the investigator will use ELISA based test system intended for the quantitative measurement of total and free testosterone for patients of both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women (primigravidas) at third trimester i.e. 28-40 weeks.
2. Age between 20 and 35 years old.
3. Live fetus.
4. Having no history of pregestational hypertension.
5. Having no history of diseases associated with hormone disorders (thyroid gland disorders, DM, hyperprolactinemia or polycystic ovary syndrome).
6. During their pregnancy they did not receive antihypertensive medications.
7. Nonsmoker.

Exclusion Criteria:

* 1- First and second trimester pregnant women. 2- Women younger than 20 years old and older than 35 years old 3- Intrauterine fetal death. 4- History of pregestational hypertension. 5- History of hormonal disorders (thyroid gland disorders and hyperprolactinemia).

  6- Smoker. 7- Polycystic ovary syndrome. 8- Signs or symptoms of hyper-androgenism (hirsutism, acne, oily skin, etc.). 9- Diabetes mellitus. 10- Drug use except ordinary supplementation (iron, folic acid).

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Study Site:
  Ain Shams University Maternity Hospital
  Study Design:
  This study is a case control study.
  Study Population:
  Patients will be divided into two groups:
  Case group:
  This group will include forty (40) preeclamptic patients at the third trimester (28-40 weeks) admitted at Ain Shams University Maternity Hospital.
  Control group:
  This group will include forty (40) normotensive pregnant women at term admitted at Ain Shams University Maternity Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Total and free testosterone level | 9 months
  Higher in preeclamptic patients than normal pregnant ladies

CONTACTS AND LOCATIONS:
Overall Officials: Noha H Rabei, Professor of Obs&Gyn, Study Chair — Ain Shams Maternity Hospital; Malames M Faisal, Lecturer of Obs&Gyna, Study Director — Ain Shams Maternity Hospital; Hoda E Abd elwahab, Fellow of medical tests, Study Director — Ain Shams Hospitals
Locations (1):
- Ain Shams Maternity Hospital-Faculty of Medicine- Ain Shams University, Cairo Governorate, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] https://www.ncbi.nlm.nih.gov/pubmed/12746983